CLINICAL TRIAL: NCT03725839
Title: The Evaluation of an Interface for the Treatment of Obstructive Sleep Apnea (OSA)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Fisher and Paykel Healthcare (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CIA-249
Record Dates: First submitted 2018-10-28; First posted 2018-10-31 (Actual); Last update posted 2020-02-28 (Actual); Status verified 2020-02

CONDITIONS: Sleep Disordered Breathing; Obstructive Sleep Apnea
MeSH Terms: conditions — Sleep Apnea Syndromes; Sleep Apnea, Obstructive

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Arm (Experimental): F&P Interface will be used by OSA participants in-home for 2 weeks.
  Interventions: Device: F&P Interface

INTERVENTIONS:
Device: F&P Interface — F&P Interface to be used for OSA therapy

SUMMARY:
This investigation is designed to evaluate the performance as well as the patients overall acceptance of the interface.

DETAILED DESCRIPTION:
A minimum of 40 OSA participants who currently use CPAP will be recruited for the trial. Participant will be in the trial for three weeks- first week will be a collection of Positive Airway Pressure baseline data on participant's usual interface. The participant will then use the trial interface in-home for 2 weeks. There is also an option of a six month extension if the participant wish to continue on the trial interface.

ELIGIBILITY:
Inclusion Criteria:

* Adult (18+ years of age)
* Able to give written consent
* AHI ≥ 5 on diagnostic night
* Either prescribed APAP, CPAP or Bi-level PAP for OSA

Exclusion Criteria:

* Inability to give written consent
* Anatomical or physiological conditions making PAP therapy inappropriate
* Commercial drivers who are investigated by New Zealand Transport Agency (NZTA)
* Current diagnosis of respiratory disease or CO2 retention
* Pregnant or may think they are pregnant.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 33 (Actual)
Dates: Start 2018-11-05 (Actual); Primary Completion 2019-11-30 (Actual); Study Completion 2019-11-30 (Actual)

PRIMARY OUTCOMES:
Trial Mask usability | 14 ± 4 days in home
  Questionnaire on ease-of-use (very easy to very difficult) Subjective
Trial mask Performance | 14 ± 4 days in home
  Questionnaire on performance (very good to very poor)- Subjective

SECONDARY OUTCOMES:
Trial mask Reliability | 5 months and 2 weeks in home
  Questionnaire on reliability - Subjective
Trial mask performance measured in L/min | 14 ± 4 days in home
  Objective leak data from PAP device

CONTACTS AND LOCATIONS:
Overall Officials: Bhavi Ogra, Principal Investigator — Clinical Manager
Locations (3):
- New Zealand (3):
  - Hawkes Bay Fallen Soldiers' Memorial Hospital, Hastings, Hawkes Bay
  - Fisher & Paykel Healthcare, Auckland
  - Well Sleep, Wellington